CLINICAL TRIAL: NCT00494481
Title: A Phase II, Double-blind, Placebo Controlled, Randomized Study to Assess the Efficacy and Safety of ZD6474 in Combination With Docetaxel (Taxotere™) vs Docetaxel Alone as 2nd Line Treatment for Advanced Breast Cancer (ABC).
Brief Title: E3 Breast Cancer Taxotere Combination
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4200C00046; 2005-003592-20 (EudraCT Number)
Record Dates: First submitted 2007-06-28; First posted 2007-06-29 (Estimated); Results first posted 2011-05-24 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-08

CONDITIONS: Advanced Breast Cancer
Keywords: Zactima
MeSH Terms: interventions — vandetanib; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Docetaxel + placebo vandetanib
  Interventions: Drug: Docetaxel
- 2 (Experimental): Vandetanib + Docetaxel
  Interventions: Drug: Vandetanib (ZD6474); Drug: Docetaxel

INTERVENTIONS:
Drug: Vandetanib (ZD6474) — once daily oral dose
  Other Names: ZACTIMA™
  Arms: 2
Drug: Docetaxel — intravenous infusion
  Other Names: Taxotere®

SUMMARY:
To assess the efficacy of ZD6474 in combination with docetaxel in the treatment of ABC using the progression event count methodology

ELIGIBILITY:
Inclusion Criteria:

* Females with histological/cytological confirmation of breast cancer.
* Subjects with a measurable lesion or bone lesions

Exclusion Criteria:

* Previous radiotherapy within 6 weeks
* Significant cardiac events, arrhythmias or other cardiac conditions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2006-01; Primary Completion 2007-06 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (12):
- Hungary (2):
  - Research Site, Budapest
  - Research Site, Pécs
- South Africa (3):
  - Research SIte, Bloemfontein
  - Research Site, Cape Town
  - Research Site, Observatory
- Spain (3):
  - Research Site, Barakaldo
  - Research SIte, Lleida
  - Research Site, Zaragoza
- Sweden (3):
  - Research Site, Umeå
  - Research Site, Uppsala
  - Research Site, Västerås
- Research Site, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient randomised 03 February 2006, last patient randomised 25 April 2007, data cut off data 23 June 2007
Groups:
- Vandetanib Plus Docetaxel: vandetanib 100 mg plus docetaxel
- Placebo Plus Docetaxel: placebo plus docetaxel
Period: Overall Study
Arm/Group | Vandetanib Plus Docetaxel | Placebo Plus Docetaxel
Started | 35 (randomised patients) | 29 (randomised patients)
Completed | 6 (ongoing study treatment at data cut-off) | 5 (ongoing study treatment at data cut-off)
Not Completed | 29 | 24
Not completed — Condition under investigation worsened | 11 | 13
Not completed — Adverse Event | 15 | 11
Not completed — Other | 1 | 0
Not completed — Never received IP | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vandetanib Plus Docetaxel | Placebo Plus Docetaxel | Total
Number analyzed (Participants) | 35 | 29 | 64
Age, Continuous [Mean (Full Range); unit: Years] | 54 [33 to 80] | 57 [39 to 74] | 55.5 [33 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 29 | 64
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With a Disease Progression Event
Description: Number of patients with objective disease progression or death (by any cause in the absence of objective progression)
Time Frame: RECIST tumour assessments carried out at screening (within 3 weeks before the 1st dose) and then as per site clinical practice until objective progression. The only additional mandatory RECIST assessment is at the point of data cut-off
Measure: Number; unit: Participants
Arm/Group | Vandetanib Plus Docetaxel | Placebo Plus Docetaxel
Number analyzed (Participants) | 35 | 29
Participants | 24 | 18

ADVERSE EVENTS:
Arm/Group | Vandetanib Plus Docetaxel | Placebo Plus Docetaxel
Serious Adverse Events (participants affected / at risk) | 14/33 | 12/29
Other Adverse Events (participants affected / at risk) | 33/33 | 25/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vandetanib Plus Docetaxel (N=33) | Placebo Plus Docetaxel (N=29)
Neutropenia (Blood and lymphatic system disorders) | 4 | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 | 1
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Keratitis (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Neutropenic Sepsis (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 1 | 0
Pharyngitis Streptococcal (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Tooth Abscess (Infections and infestations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Vocal Cord Paralysis (Nervous system disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis Exfoliative (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Papular (Skin and subcutaneous tissue disorders) | 1 | 0
Toxic Epidermal Necrolysis (Skin and subcutaneous tissue disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vandetanib Plus Docetaxel (N=33) | Placebo Plus Docetaxel (N=29)
Neutropenia (Blood and lymphatic system disorders) | 15 | 13
Leukopenia (Blood and lymphatic system disorders) | 10 | 8
Anaemia (Blood and lymphatic system disorders) | 6 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 | 0
Lymphopenia (Blood and lymphatic system disorders) | 3 | 2
Agranulocytosis (Blood and lymphatic system disorders) | 2 | 2
Vertigo (Ear and labyrinth disorders) | 2 | 1
Lacrimation Increased (Eye disorders) | 2 | 7
Conjunctivitis (Eye disorders) | 2 | 3
Vision Blurred (Eye disorders) | 0 | 2
Stomatitis (Gastrointestinal disorders) | 16 | 12
Diarrhoea (Gastrointestinal disorders) | 13 | 12
Nausea (Gastrointestinal disorders) | 9 | 10
Abdominal Pain (Gastrointestinal disorders) | 6 | 5
Vomiting (Gastrointestinal disorders) | 3 | 6
Constipation (Gastrointestinal disorders) | 5 | 2
Dry Mouth (Gastrointestinal disorders) | 4 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 3 | 3
Flatulence (Gastrointestinal disorders) | 2 | 1
Gastritis (Gastrointestinal disorders) | 2 | 2
Mouth Ulceration (Gastrointestinal disorders) | 0 | 2
Odynophagia (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 11 | 7
Asthenia (General disorders) | 3 | 8
Oedema Peripheral (General disorders) | 7 | 6
Pyrexia (General disorders) | 5 | 3
Face Oedema (General disorders) | 1 | 2
Influenza Like Illness (General disorders) | 1 | 2
Malaise (General disorders) | 2 | 0
Performance Status Decreased (General disorders) | 2 | 0
Pharyngitis (Infections and infestations) | 2 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 3
Herpes Zoster (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 2 | 1
Oral Candidiasis (Infections and infestations) | 1 | 2
Urinary Tract Infection (Infections and infestations) | 2 | 0
Chemical Eye Injury (Injury, poisoning and procedural complications) | 2 | 2
Weight Decreased (Injury, poisoning and procedural complications) | 3 | 2
Alanine Aminotransferase Increased (Injury, poisoning and procedural complications) | 2 | 2
Aspartate Aminotransferase Increased (Injury, poisoning and procedural complications) | 2 | 2
Blood Alkaline Phosphatase Increased (Injury, poisoning and procedural complications) | 2 | 1
Anorexia (Metabolism and nutrition disorders) | 7 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 9
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Paraesthesia (Nervous system disorders) | 4 | 9
Peripheral Sensory Neuropathy (Nervous system disorders) | 6 | 3
Dysgeusia (Nervous system disorders) | 5 | 4
Headache (Nervous system disorders) | 4 | 4
Hypoaesthesia (Nervous system disorders) | 4 | 3
Dizziness (Nervous system disorders) | 3 | 2
Lethargy (Nervous system disorders) | 3 | 3
Neurotoxicity (Nervous system disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 3 | 2
Depression (Psychiatric disorders) | 2 | 1
Dysuria (Renal and urinary disorders) | 2 | 1
Vaginal Discharge (Reproductive system and breast disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 17 | 11
Erythema (Skin and subcutaneous tissue disorders) | 7 | 4
Onycholysis (Skin and subcutaneous tissue disorders) | 6 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 5 | 5
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 5 | 0
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 2 | 5
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 3 | 4
Acne (Skin and subcutaneous tissue disorders) | 3 | 1
Nail Discolouration (Skin and subcutaneous tissue disorders) | 3 | 0
Nail Pigmentation (Skin and subcutaneous tissue disorders) | 3 | 3
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 3 | 0
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1 | 3
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 | 3
Nail Disorder (Skin and subcutaneous tissue disorders) | 2 | 2
Pigmentation Disorder (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Rash Pruritic (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 5 | 0
Flushing (Vascular disorders) | 2 | 2
Hot Flush (Vascular disorders) | 0 | 2
Lymphoedema (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.